CLINICAL TRIAL: NCT06039904
Title: Comparison Between Natural Rubber Knee Support and Sponge Knee Support on the Protection of Knee Joint: A Crossover Randomized Controlled Study Among Patients With Bleeding Disorders
Brief Title: Protection of Knee Joints in Bleeding Disorder Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Nongnuch Sirachainan, Prof, Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: COA.MURA2021/292
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Bleeding Disorder; Knee Injuries; Hemophilia
MeSH Terms: conditions — Hemostatic Disorders; Knee Injuries; Hemophilia A

STUDY DESIGN:
Intervention Model Description: Randomized crossover trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A was first assigned to Treatment I of natural rubber knee support followed by Treatment II of sponge knee support
  Interventions: Device: Natural rubber knee support
- Arm B (Experimental): Arm B was first assigned to Treatment II of sponge knee support followed by Treatment I of natural rubber knee support
  Interventions: Device: Sponge knee support

INTERVENTIONS:
Device: Natural rubber knee support — The knee support comprised two parts, the support body and the protective cushion. Which were categorized into four sizes, S, M, L and XL according to widths and lengths, as follows: size S, 8x17 cm; size M, 10x19 cm; size L, 12x24 cm; and size XL, 14x28 cm. The support body was made of stretchable natural cotton fabrics, which were comfortable, breathable, washable, less irritant and flexible. Similarly, the protective cushion was classified into four sizes: S, M, L and XL with diameters (based on the patellar diameters) of 5, 6, 7 and 8 cm, respectively. Cushions were made from either natural rubber and inserted at the front of the support body (to cover the patellar).
  Other Names: Sponge knee support
  Arms: Arm A
Device: Sponge knee support — The knee support comprised two parts, the support body and the protective cushion. Which were categorized into four sizes, S, M, L and XL according to widths and lengths, as follows: size S, 8x17 cm; size M, 10x19 cm; size L, 12x24 cm; and size XL, 14x28 cm. The support body was made of stretchable natural cotton fabrics, which were comfortable, breathable, washable, less irritant and flexible. Similarly, the protective cushion was classified into four sizes: S, M, L and XL with diameters (based on the patellar diameters) of 5, 6, 7 and 8 cm, respectively. Cushions were made from either sponge and inserted at the front of the support body (to cover the patellar).
  Arms: Arm B

SUMMARY:
INTRODUCTION Knee supports, usually made with sponge cushion, are used to protect knee joint and prevent its injury. Sponge has less elasticity and durability compared with natural rubber. To our knowledge, there has been no study regarding effectiveness of natural rubber and sponge for knee joint protection and injury prevention in children with bleeding disorders.

AIMS The study aimed to compare the effectiveness and satisfaction between natural rubber and sponge knee supports for knee joint protection among children with bleeding disorders METHODS The study had three phases: 1) measurement of compression force, 2) fabrication of knee supports, and 3) a randomized crossover trial. The supports were fabricated in 4 sizes, S, M, L, and XL. They comprised two parts: body, made from stretchable cotton; and cushion (protection part), made from either natural rubber or sponge. The trial included 8 weeks of alternatively wearing natural rubber knee support and sponge knee support with a 4-week wash-out period. Numbers of knee bleeds and satisfied users were recorded.

DETAILED DESCRIPTION:
The study employed a prospective design, conducted at the Faculty of Medicine Ramathibodi Hospital, a tertiary care hospital in Thailand, from April 2021 to September 2022; and approved by the Hospital's Committee on Human Rights Related to Research Involving Human Subjects (COA. MURA2021/292). Written informed consents were obtained from individual patients and their legal guardians. The study was divided into three phases: measurement of transmitted impact force, fabrication of knee supports, and randomized cross-over trial of natural rubber and sponge knee supports.

Phase I: Transmitted impact forces were measured using an impact tester (Model DC Power Supply GW Instek GPS-30300 and Multi-Meter Fluke DT-9208a). Three types of knee support samples, size 30 x 30 x 1 cm (W x L x H), were prepared: with no barrier, with natural rubber cushion, and with sponge cushion and tested. The test was performed using the same force in the ballistic pendulum test (1 kg momentum ball with a radius of 50 cm). The test was repeated three times, and the average results were recorded as force (Newton) and time (sec) after the sphere hit the receptive sensor. Natural rubber used in this study was made from natural rubber and polymer (Patent ID 74814).

Phase II: Knee supports were designed and fabricated in various sizes. Three measurements, knee circumferences, patella sizes, and knee heights, were taken from 20 Thai children aged between 9 months and 10 years and having body weights within the 50th to 75th percentile. The knee support comprised two parts, the support body and the protective cushion. The width of the support body was derived from half of the knee circumference, and the length was taken from 80% of the knee height, measured from knee to medial malleolus. From those measurements, final knee supports were categorized into four sizes, S, M, L and XL according to widths and lengths, as follows: size S, 8x17 cm; size M, 10x19 cm; size L, 12x24 cm; and size XL, 14x28 cm. The support body was made of stretchable natural cotton fabrics, which were comfortable, breathable, washable, less irritant and flexible.22 Similarly, the protective cushion was classified into four sizes: S, M, L and XL with diameters (based on the patellar diameters) of 5, 6, 7 and 8 cm, respectively. Cushions were made from either natural rubber or sponge and inserted at the front of the support body (to cover the patellar). As a result, natural rubber and sponge knee supports were fabricated, and they both had similar external appearance.

Phase III: A randomized cross-over trial using natural rubber and sponge knee supports was conducted among patients with bleeding disorders. The patients were divided into two groups, A and B, by computer-generated randomization sequence using a box of ten. A total of 44 patients were enrolled with 21 in Group A and the other 23 in Group B. Later, two patients in Group A were excluded due to loss of follow-ups. Therefore, the final number of patients in the study was 42 with 19 in Group A and 23 in Group B. Group A was first assigned to Treatment I of natural rubber knee support followed by Treatment II of sponge knee support, while Group B was first assigned to Treatment II followed by Treatment I. Patients were advised to use the supports during physical activities; for example, walking and crawling among toddlers and playing sports among school-aged children. Each treatment covered a period of eight weeks, with four weeks of wash-out period of cross-over from the first treatment to the second. Survey data on demographics, number of bleeds, types of bleeding (extraarticular or intraarticular), and user's satisfaction were collected. User's compliance and bleeding data, including severity and activity when injury occurred, were collected weekly using freeware application, online electronic form, or direct telephone contact. Satisfaction survey was conducted following the Client Satisfaction with Device module of Orthotics and Prosthetic User' Survey (CSD-OPUS)24 with Thai translation. The survey consisted of nine aspects: fitting well, weight, comfort, ease to use, attractiveness, durability, irritation, pain, and overall satisfaction. Patients aged >7 years and all parents were included in the survey, sent to them in electronic format, twice; i.e., at the end of the two treatments. Scores were graded in absolutely agree, agree, disagree, and absolutely disagree. At the end of the second treatment, parents of both groups were asked to choose either the knee support of Treatment I or Treatment II as a preference.

Patients The inclusion criteria were bleeding disorder patients, aged 9 months to 12 years old, with written consents The enrolled patients had no coexisting diseases affecting their activities, or bleeding episodes two weeks before the study. Children or parents who were not able to continue the study until the end were excluded.

ELIGIBILITY:
Inclusion Criteria:

* bleeding disorder patients, aged 9 months to 12 years old, with written consents

Exclusion Criteria:

* coexisting diseases affecting their activities, or bleeding episodes two weeks before the study

Ages: 9 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Number of knee bleeding | 8 weeks
  Number of intra and extraarticular knee bleedings

CONTACTS AND LOCATIONS:
Locations (1):
- Supicha Maneekhiew, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No